CLINICAL TRIAL: NCT05855239
Title: Quantification of Hepatic Steatosis in Patients With Fatty Liver Disease Using Attenuation Imaging With Different Ultrasound Frequency
Brief Title: Quantification of Hepatic Steatosis With Different Ultrasound Frequency
Status: Active, not recruiting | Type: Observational
Sponsor: Jong Keon Jang (Other)
Collaborators: Canon Medical Systems, Korea (Unknown)
Responsible Party: Sponsor-Investigator, Jong Keon Jang, Assistant Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: ATI_Freq_01
Record Dates: First submitted 2023-04-29; First posted 2023-05-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Fatty Liver; Fatty Liver, Nonalcoholic; Ultrasound
Keywords: Hepatic steatosis; Quantification; Ultrasound; Attenuation coefficient
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is: (1) to compare the feasibility (technical successes rate and reliability) in measuring attenuation coefficient between two different frequencies (3MHz, 4MHz) of ultrasound beam; (2) to evaluate and compare the diagnostic performance of attenuation coefficient for steatosis using two different frequencies (3MHz, 4MHz) of ultrasound beam by comparison with the pathologic results acquired by liver biopsy or surgery.

DETAILED DESCRIPTION:
Investigators measure the distance between the skin and liver capsule on B-mod images.

Investigators place a region of interest (ROI) avoiding reverberation artifacts and acquire attenuation coefficient for five times.

For participants who require a liver biopsy, investigators try to target the same area in the liver, where ROI was placed.

Investigators evaluate hepatic steatosis, lobular inflammation, and fibrosis of tissue of the liver using a scoring system suggested by Nonalcoholic Steatohepatitis Clinical Research Network.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are candidates for liver donation and scheduled liver biopsies for assessment of hepatic steatosis
* Participants suspected of nonalcoholic fatty liver disease and scheduled for liver biopsy or surgery

Exclusion Criteria:

* Participants with a BMI of less than 23
* Participants underwent liver transplantation or right hepatectomy
* Participants who have a large mass in the right liver
* Participants who have a bleeding tendency (platelet count < 80000, prothrombin time and international normalized ratio > 1.5)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at risk of fatty liver disease
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Attenuation coefficient (3MHz vs. 4MHz) in attenuating imaging | During procedure
  dB/cm/MHz
Percentage of fat within hepatocyte in pathological specimen | During procedure
  S0 (<5%), S1(5%~33%), S2(34%~66%), and S3 (>66%)

CONTACTS AND LOCATIONS:
Overall Officials: JongKeon Jang, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, P’ungnap-tong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
No plan to share data with another researcher